CLINICAL TRIAL: NCT05237180
Title: Evaluation of the Effect of a Spatial Localization Training Program on Auditory Comprehension in Noise in Bi-implanted Subjects With Post-lingual Deafness
Brief Title: Evaluation of the Effect of a Spatial Localization Training Program on Auditory Comprehension
Acronym: CAudiBruit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/CHU/32
Record Dates: First submitted 2022-01-10; First posted 2022-02-14 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-01

CONDITIONS: Hearing Loss, Cochlear
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient group (Experimental): 8 training sessions on spatial localisation
  Interventions: Other: spatial localisation training
- control croup (No Intervention): Non training sessions

INTERVENTIONS:
Other: spatial localisation training — 8 spatial localization training sessions MBAA and SSQ tests before and after training sessions.
  Arms: patient group

SUMMARY:
Hearing comprehension under complex listening conditions is considered to be the central complaint of everyday life for patients with cochlear implants. Localization is one of the cues for listening comprehension. However, only few studies have investigated the effect of spatial localization training on listening comprehension performance in noise. None of these studies correspond to the desire to purpose training by speech therapists while using affordable equipment.

The main objective of this study is to evaluate the effect of a spatial localization training protocol in cochlear bi-implanted subjects with post-lingual deafness on their ability to understand in noise.

2 groups of 10 subjects each will be recruited: a patient group and a control group. The patient group will undergo 8 sessions of spatial localization rehabilitation lasting an average of 45 minutes each.

After this programme, the pre-test and post- test results obtained will be compared.

ELIGIBILITY:
Inclusion Criteria:

* post-lingual deafness
* implanted bilaterally for at least 1 year
* score ≥ 70 at LAFON scale
* score ≥ 70 at MBAA scale
* score ≥ 5/9 at CAP scale
* good command of the French language
* accepts to participate in the study

Exclusion Criteria:

* do not realize speech reeducation (spatial localisation and speech perception) during the study
* no change in setting of cochlear implants

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Change of Hearing comprehension performance in noise | 10 weeks after inclusion
  MBAA (Marginal Benefic from Acoustical Amplification) scale. Minimal score = 0 and maximal score =540. minimum score means that the patient is unable to repeat phrases and maximal score means that the patient is able to repeats all phrases.
Change of Hearing comprehension performance in noise | 10 weeks after inclusion
  15iSSQ (New 15 items Speech Spatial and qualities of hearing Scale Shoirt Form). Minimum score =0 and maximal score = 150. maximal score means that the patient has a good quality of life and minimum score means that his quality of life is bad.
  It is a qualitative evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Justine MAISSON, Principal Investigator — GCS CRCSI
Locations (1):
- Gcs Crcsi, Sainte-Clotilde, Reunion

IPD SHARING:
Plan to Share IPD: No